CLINICAL TRIAL: NCT07084363
Title: Quantitative Versus qUAlitative NeuromoniToring of neUroMuscular Block for Non-cardiothoracic Surgery (The QUANTUM Trial): Single-center Cluster Randomized Multiple Crossover Trial
Brief Title: Quantitative Versus qUAlitative NeuromoniToring of neUroMuscular Block for Non-cardiothoracic Surgery
Acronym: QUANTUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mehmet Turan, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-25-0337
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Neuromuscular Block, Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Intervention Model Description: Designated operating rooms of the hospital will be cluster randomized in this study. For each week of the 24-week trial, the designated operating rooms will be randomized to either quantitative or qualitative TOF monitoring.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Quantitative monitoring (Experimental)
  Interventions: Device: Quantitative monitoring
- Qualitative monitoring (Active Comparator)
  Interventions: Other: Qualitative monitoring

INTERVENTIONS:
Device: Quantitative monitoring — The TetraGraph TOF monitor will be used to quantitatively assess the TOF-ratio. Quantitative monitoring includes objective measurement of the TOF-ratio, as defined by the ratio between the first and the fourth muscular responses and is quantified by acceleromyography. A TOF twitch response ratio equal or greater to 95% (TOF0.95) will be targeted prior to extubation. If TOF0.95 is not reached within 10 min of administering the initial dose of the respective reversal agent, redosing is recommended.
  Arms: Quantitative monitoring
Other: Qualitative monitoring — Clinicians will assess the TOF-ratio. Qualitative monitoring includes subjective assessment of the count and the amplitude of the muscular responses related to neuromuscular block depth. A TOF twitch response count of 4 similarly strong twitches will be targeted prior to extubation. If 4 similarly strong TOF twitch responses are not reached within 10 min of administering the initial dose of the respective reversal agent, redosing is recommended.
  Arms: Qualitative monitoring

SUMMARY:
The purpose of this study is to assess the effect of quantitative block monitoring versus less expensive qualitative monitoring treatment effects on the lowest SpO2/FiO2 ratio in the PACU. The results will be incorporated into an enhanced recovery pathway for surgical patients.

ELIGIBILITY:
Inclusion criteria:

* Patient age ≥ 18 years old;
* General anesthesia with endotracheal intubation;
* Neuromuscular block with rocuronium.

Exclusion criteria:

* Intubation before induction of anesthesia;
* Critically ill patients admitted from the ICU;
* Emergency cases;
* Non-intubated patients;
* Patients who will not be paralyzed through the surgery (spine).
* Patients with an implanted electronic device (e.g. cardiac pacemaker)
* Patients with allergies to adhesive
* Patients with pre-existing neuromuscular disease (e.g. Myasthenia Gravis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1032 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
lowest SpO2/FiO2 ratio in the PACU (constant for at least 10 minutes) | During the time in PACU (about 30 minutes to 6 hours)

SECONDARY OUTCOMES:
Collapsed composite (any vs none) of postoperative pulmonary complications | During length of hospital stay (about 1 day to a week)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Turan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No